CLINICAL TRIAL: NCT06856707
Title: MIRA Surgical System Registry Study (MIRA Registry)
Brief Title: MIRA Registry Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Virtual Incision Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 110-002103
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Colon Procedures; Bowel Resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Surgical: Patients undergoing surgery with the MIRA Surgical System
  Interventions: Device: Use of the MIRA Surgical System during surgery

INTERVENTIONS:
Device: Use of the MIRA Surgical System during surgery — Use of the MIRA Surgical System to perform robotically assisted colorectal surgery.
  Other Names: Robotically Assisted Surgery

SUMMARY:
The purpose of the MIRA Surgical System Registry is to accumulate and evaluate real world evidence experience as part of post-market surveillance using the MIRA Surgical System.

The studies primary goals are to:

* To evaluate the performance of the MIRA Surgical System
* To evaluate the Device Safety profile

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery using the MIRA Surgical System
* Subject is able to provide informed consent
* Subject is available for post operative follow up visit through 30 days

Exclusion Criteria:

* Has or is participating in another clinical trial which may confound study results
* In the opinion of the investigator, patient is not likely to complete post-operative care and/or return for standard follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients indicated for minimally invasive surgery using the MIRA Surgical System.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-05-28 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Performance of MIRA Surgical System | From time of procedure through completion of the surgical procedure
  Successful completion of the surgical procedure using the MIRA Surgical System without conversion to open surgery (Yes/No).
Device Safety | From time of surgery using the MIRA Surgical System through 30 days following surgical procedure
  Incidence of Device related adverse events and Unanticipated Device Effects

CONTACTS AND LOCATIONS:
Overall Officials: Piet Hinoul, M.D., Study Chair — Virtual Incision Corporation
Locations (1):
- Bryan Medical Center, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Study design is to evaluate cumulative database of all patients who have undergone surgery using the MIRA Surgical System.